CLINICAL TRIAL: NCT04625517
Title: Performance of Contrast-Enhanced Spectral Mammography to Assess Neoadjuvant Chemotherapy Response (CEDM)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Basak Dogan, MD, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2019-0529
Record Dates: First submitted 2020-11-04; First posted 2020-11-12 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: mammography; contrast enhanced spectral mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Breast cancer patients (Experimental): Patients with ipsilateral intact biopsy-proven breast cancer
  Interventions: Procedure: Digital Mammography; Drug: Low Osmolar Contrast Material, 300-399 Mg/Ml Iodine Concentration, Per Ml

INTERVENTIONS:
Procedure: Digital Mammography — Digital Mammography enhanced with an iodinated contrast agent
Drug: Low Osmolar Contrast Material, 300-399 Mg/Ml Iodine Concentration, Per Ml — Injection of low osmolar contrast material during the digital mammography exam

SUMMARY:
This study is designed to investigate the diagnostic accuracy of Contrast Enhanced Spectral Mammography (CEDM) in predicting early neoadjuvant therapy response and pathologic complete response (pCR) compared to mammography.

Patients diagnosed with invasive breast cancer with available mammography and ultrasound imaging are eligible for the study.

Eligible patients will be imaged at baseline (before initiation of neoadjuvant chemotherapy or endocrine therapy), early (2-4 cycles of neoadjuvant therapy) and late (after completion of neoadjuvant chemotherapy or endocrine therapy) timepoints with mammography. CEDM will be done within 2 weeks of the specified timepoint. Additionally, a survey of subject experience with CEDM and other pre-operative imaging will be collected after CEDM is performed.

DETAILED DESCRIPTION:
The use of neoadjuvant systemic therapy in the treatment of breast cancer patients is increasing beyond the scope of locally advanced disease. Imaging provides important information in assessing response to therapy as a complement to conventional tumor measurements via physical examination. Tumor response to neoadjuvant therapy can also provide prognostic information. The attainment of pCR after completion of neoadjuvant therapy and surgical resection is associated with improved disease-free survival. This correlation is especially strong for Triple-receptor negative and human epidermal growth factor receptor 2 (HER-2) positive breast cancer. Studies of neoadjuvant therapy have used a variety of methods for assessing tumor response. Currently, there are no established clinical practice guidelines for how best to assess tumor response to neoadjuvant therapy. Typically, patients undergo conventional breast imaging such as mammography and ultrasonography (US) and physical examination, and dynamic contrast-enhanced breast magnetic resonance imaging (DCR-MRI) in selected cases.

Contrast Enhanced Digital Mammography (CEDM) is a novel imaging technique, which allows digital mammography to be used with contrast enhancement to depict cancers that would otherwise be occult on standard unenhanced mammography. CEDM is performed with and without intravenous iodine contrast, using the dual energy subtraction technique. Compared with mammography and US, CEDM improves the sensitivity for breast cancer detection without decreasing specificity. CEDM digital detector has higher spatial resolution than MRI, revealing details that are approximately 10 times better. In contrast to the rapid washout in MRI, enhancement on CEDM in fact persists for at least 10 min after contrast agent infusion. Today CEDM is available commercially for clinical use. It is estimated that over 200,000 CEDM examinations have been performed to date in both research and clinical settings. CEDM costs significantly less compared to MRI. Furthermore, longer time delays between contrast injection and CEDM exposure could result in stronger enhancement and hence better visibility compared to MRI, especially given the much higher spatial resolution of digital mammography. It is unknown whether CEDM can improve the sensitivity of mammography in the early assessment of neoadjuvant therapy response. We hypothesize that CEDM is superior to mammography and ultrasound in assessing early response, and pre-surgical residual cancer after neoadjuvant therapy, and when performed, non-inferior to MRI in assessing the residual disease using the metrics of pCR and residual cancer burden (RCB).

ELIGIBILITY:
Inclusion Criteria:

* Ipsilateral intact biopsy-proven breast cancer clinical stage T1-T4 (by imaging)
* Available mammography and ultrasound imaging of the existing index cancer, with orthogonal measurements
* Prior history of ipsilateral or contralateral breast cancer, presenting with a new primary or recurrent disease
* Patients who were determined to be candidates for either neoadjuvant chemotherapy or neoadjuvant endocrine therapy by the treating physician
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for days following completion of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* History of ipsilateral mastectomy
* Women who already started neoadjuvant chemotherapy or endocrine therapy
* Woman who may be pregnant or nursing an infant
* Prior history of anaphylactic or anaphylactoid reaction to any contrast.
* Prior allergy to iodine or iodinated contrast.
* Impaired renal function measured by estimated glomerular filtration rate (eGFR) < 60 milliliters per minute.
* Patients with known distant metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Basak Dogan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Breast Cancer Patients
Started | 6
Completed | 3
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Predicting pCR (Pathologic Complete Response) for CEDM
Description: Sensitivities in predicting pCR will be calculated for CEDM and measured as AUC
Time Frame: 4 to 6 months from initiation of neoadjuvant therapy until final surgery
Population: The number of participants with outcomes in our trial was limited to only three. Furthermore, none of the patients had pCR -hence none of the cases have the reference standard needed to calculate this parameter (sensitivity).
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 0

2. Primary Outcome: Sensitivity of Predicting pCR (Pathologic Complete Response) for Mammography
Description: Sensitivities in predicting pCR will be calculated for mammography measured as AUC
Time Frame: 4 to 6 months from initiation of neoadjuvant therapy until final surgery
Population: as for outcome 1
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 0

3. Primary Outcome: Specificity of Predicting pCR (Pathologic Complete Response) for CEDM
Description: Specificity of predicting pCR will be calculated for CEDM and measured as AUC
Time Frame: 4 to 6 months from initiation of neoadjuvant therapy until final surgery
Population: The number of participants with outcomes in our trial was limited to only three. Furthermore, none of the patients had pCR -hence none of the cases have the reference standard needed to calculate this parameter (specificity).
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 0

4. Primary Outcome: Specificity of Predicting pCR (Pathologic Complete Response) for Mammography
Description: Specificity of predicting pCR will be calculated for mammography and measured as AUC
Time Frame: 4 to 6 months from initiation of neoadjuvant therapy until final surgery
Population: as for outcome 3
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 0

5. Primary Outcome: Diagnostic Accuracy of Contrast-enhanced Mammography in Assessing pCR or Non Response
Description: ROC analysis will be used to assess the diagnostic performance of CEDM. The Area under the receiver operating characteristic (ROC) curve (AUC) will be compared. A leave-one-out cross validation algorithm will be used to reduce bias from overfitting.
Time Frame: 4 to 6 months from initiation of neoadjuvant therapy until final surgery
Population: The number of participants with outcomes in our trial was limited to only three. Furthermore, none of the patients had pCR - hence absence of reference standard end point precludes this assessment.
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 0

6. Primary Outcome: Correlation of Residual Tumor Size With Pathologic Size
Description: Spearman's rank correlation will be used to measure the association between final pathologic and imaging tumor size
Time Frame: 4 to 6 months from initiation of neoadjuvant therapy until final surgery
Population: The number of participants with outcomes in our trial was limited to only three. Furthermore, none of the patients had pCR -hence none of the cases have the reference standard needed to calculate this parameter.
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: At least 30 minutes after contrast administration
Description: Only contrast-specific side effects were collected for this study
Arm/Group | Breast Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT04625517/Prot_SAP_000.pdf